CLINICAL TRIAL: NCT00551148
Title: PD 0200390 Dose-ranging Trial: A Randomized, Double-blind, Placebo-controlled, 5-way Crossover, Multicenter Polysomnography Trial of PD 0200390 in Adults With Primary Insomnia
Brief Title: A Dose-ranging, Multicenter Polysomnography Trial of PD 0200390 in Adults With Primary Insomnia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: A4251068
Record Dates: First submitted 2007-10-27; First posted 2007-10-30 (Estimated); Last update posted 2012-07-25 (Estimated); Status verified 2012-07

CONDITIONS: Primary Insomnia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — (1-aminomethyl-3,4-dimethylcyclopentyl)acetic acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- 15 mg (Experimental)
  Interventions: Drug: PD 0200390
- 30 mg (Experimental)
  Interventions: Drug: PD 0200390
- 5 mg (Experimental)
  Interventions: Drug: PD 0200390
- 60 mg (Experimental)
  Interventions: Drug: PD 0200390
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: PD 0200390 — oral 15 mg dose on 2 consecutive nights. This is one of 5 treatment doses administered one week apart for 5 consecutive weeks.
  Arms: 15 mg
Drug: PD 0200390 — oral 30 mg dose on 2 consecutive nights. This is one of 5 treatment doses administered one week apart for 5 consecutive weeks.
  Arms: 30 mg
Drug: PD 0200390 — oral 5 mg dose on 2 consecutive nights. This is one of 5 treatment doses administered one week apart for 5 consecutive weeks.
  Arms: 5 mg
Drug: PD 0200390 — oral 60 mg dose on 2 consecutive nights. This is one of 5 treatment doses administered one week apart for 5 consecutive weeks.
  Arms: 60 mg
Other: Placebo — oral placebo mg dose on 2 consecutive nights. This is one of 5 treatment doses administered one week apart for 5 consecutive weeks.
  Arms: Placebo

SUMMARY:
The purpose of this study is to further explore an effective dose range of PD0200390 for the treatment of patients with insomnia.

ELIGIBILITY:
Inclusion Criteria:

3 month history of Primary Insomnia (DSM-IV criteria)

Self report sleep criteria for at least 3 nights per week in past month;

sWASO (subjective wake after sleep onset) equal or greater than 60 mins

sLSO (subjective latency to sleep onset) equal or greater than 45 minutes

TST less than or equal to 6.5 hrs

Maintain normal daytime-awake, nighttime-sleep schedule

PSG sleep criteria of mean WASO equal or greater than 60 mins calculated on 2 PSG screening nights

TST between 3 to 7 hrs on 2 PSG screening nights

Mean LPS (latency to persistent sleep) equal or greater than 20 mins calculated on 2 PSG screening nights

Exclusion Criteria:

Comorbid psychiatric disease or disorders

History or presence of breathing-related disorders

Multivariable Apnea risk index (MAP) equal or greater than 0.5 at screening

History or presence of medical or neurological condition interfering with sleep

Current use of know psychotropic effect medications

Excessive caffeine use

Use of alcohol as a sleep aid or more than 2 standard drinks/day

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 92 (Actual)
Dates: Start 2007-10; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
Dose-response relationship of PD 200390 on wake after sleep onset (WASO) in subjects with primary insomnia as determined by Polysomnography | weekly

SECONDARY OUTCOMES:
Subjective assessments of wake after sleep onset (sWASO), latency to sleep onset (LSO), number of awakenings after sleep onset (sNAASO), total sleep time (TST), and sleep quality via questionnaire. | weekly
Subjective assessment of sleep with Leeds Sleep Evaluation Questionnaire-LSEQ. | weekly
PSG efficacy assessments including number of awakenings after sleep onset (NAASO), number of arousals, total sleep time (TST), sleep efficiency (SE), total wake time (TWT) | weekly
Latency to persistent sleep (LPS) as determined by Polysomnography | weekly

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (15):
- United States (15):
  - Pfizer Investigational Site, Glendale, Arizona
  - Pfizer Investigational Site, Phenoix, Arizona
  - Pfizer Investigational Site, Phoenix, Arizona
  - Pfizer Investigational Site, Tucson, Arizona
  - Pfizer Investigational Site, San Diego, California
  - Pfizer Investigational Site, Miami, Florida
  - Pfizer Investigational Site, Naples, Florida
  - Pfizer Investigational Site, South Miami, Florida
  - Pfizer Investigational Site, Atlanta, Georgia
  - Pfizer Investigational Site, Overland Park, Kansas
  - Pfizer Investigational Site, Crestview Hills, Kentucky
  - Pfizer Investigational Site, New York, New York
  - Pfizer Investigational Site, Cary, North Carolina
  - Pfizer Investigational Site, Raleigh, North Carolina
  - Pfizer Investigational Site, Cincinnati, Ohio

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A4251068&StudyName=A%20Dose-ranging%2C%20Multicenter%20Polysomnography%20Trial%20of%20PD%200200390%20in%20Adults%20with%20Primary%20Insomnia